CLINICAL TRIAL: NCT01176357
Title: Adiponectin and Inflammatory Mediators in Mediastinal Adipose Tissues Between Patients With Coronary Artery Diseases and With Valvular Diseases
Brief Title: Adiponectin and Inflammatory Mediators in Mediastinal Adipose Tissues
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Shih-Hong Huang, Far Eastern Memorial Hospital
Other Study IDs: 96039; FEMH-96-D-003
Record Dates: First submitted 2009-02-06; First posted 2010-08-06 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2010-08

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Coronary artery disease (CAD); atherosclerosis; mediastinal adipose tissue; adiponectin, inflammatory mediators
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Adipose tissue biopsy samples from mediastinal fat, epicardial fat, subcutaneous fat in thoracic region or abdominal region and subcutaneous fat in leg were obtained soon after sternotomy or thoracotomy before the initiation of cardiopulmonary bypass.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: CABG
- 2: Valve surgery

SUMMARY:
Coronary artery disease (CAD), the most common type of heart disease, is caused by hardening of the arteries, or atherosclerosis that is an inflammatory process in which immune mechanisms interact with metabolic risk factors to initiate, propagate, and activate lesions in the arterial trees. Epidemiological studies have found that increased cardiovascular risks are associated with increased levels of inflammatory cytokines (eg, interleukin-6 [IL-6] and tumor necrosis factor-alpha[TNF-alpha]) or their hepatic product, C-reactive protein (CRP). Higher expression of interleukin-Ibeta(IL-1beta),IL-6, monocyte chemotactic protein-1 (MCP-1), and TNF-alpha were observed in epicardial adipose tissues in patients with CAD. These findings suggested that the pericoronary tissues could be a source of inflammatory mediators or act as paracrine that lead to vascular inflammation on CAD pathogenesis. However, adiponectin, a kind of adipocytokine, produced and secreted exclusively by adipose tissue, has been reported to have a variety of anti-inflammatory functions against atherosclerosis, resulting in risk reduction for incidence of CAD events. It remains unclear whether adiponectin and inflammatory mediators in mediastinal adipose tissue contribute to CAD. We therefore aim to analyze the expression of adiponectin and inflammatory mediators in mediastinal adipose tissue between patients with CAD and with valve diseases, and to correlate these parameters with clinical atherosclerotic risks, medications (statins or antiplatelet), and blood sugar.

ELIGIBILITY:
Inclusion Criteria:

* patient underwent CABG or valve surgery in our hospital will be included

Exclusion Criteria:

* liver disease
* dhronic renal insufficiency
* neoplastic diseases
* taking steroids
* congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CAD or with valve diseases proposed to have cardiac operations
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Ming Chiu, MD, PhD, Principal Investigator — FEMH
Locations (1):
- FEMH, Taipei, Taiwan